CLINICAL TRIAL: NCT04651985
Title: Effects of Eccentric Strengthening Exercises in Adults With an Achilles Tendinopathy: Predictive Validity and Responsiveness of Quantitative Musculoskeletal Ultrasound Measures
Brief Title: Responsiveness of Quantitative Musculoskeletal Ultrasound Measures on the Healing of Achilles Tendon
Status: Completed | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-9100
Record Dates: First submitted 2020-11-13; First posted 2020-12-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-11

CONDITIONS: Achilles Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Injured Achilles tendon participants who have an Achilles tendinopathy: They will do the eccentric exercise protocol and go through a series of ultrasound examination.
  Interventions: Other: Eccentric strengthening exercises of the Achilles tendon
- Healthy Achilles tendon (contralateral) of participants who have an Achilles tendinopathy: They will do the eccentric exercise protocol and go through a series of ultrasound examination.
  Interventions: Other: Eccentric strengthening exercises of the Achilles tendon

INTERVENTIONS:
Other: Eccentric strengthening exercises of the Achilles tendon — This exercise will require the completion of slow active eccentric plantar flexion exercises with the forefoot positioned over the edge of a step. These exercises will be repeated twice daily (three sets of 15 repetitions with the knee in extension and three sets of 15 repetitions with the knee in flexion) during a three-month period. The amount of loading will be calibrated and progressed on a weekly basis by the physiotherapist according the participant's perceived effort and pain intensity.

SUMMARY:
To this day, the most accepted treatment for the Achilles tendinopathy (AT) remains the exercise program to strengthen the plantar flexor muscles. The eccentric exercises protocol proposed by Alfredson is the most popular and recommended one by the rehabilitation professionals. Currently, the response to interventions is measured almost exclusively by clinical data, especially using questionnaires, since the Quantitative Ultrasound (QUS) is rarely used. In fact, the thickness of the Achilles tendon, which is generally the only measure noted when using musculoskeletal ultrasound on AT, does not allow the clinician to confirm an improvement following an eccentric exercise program if the tendon is thinner, especially in adults with chronic AT. No scientific evidence indicates whether there is an improvement in the biological integrity of the Achilles tendon following the completion of Alfredson's eccentric strengthening protocol. This is why it seems relevant to use the pre-established minimal biomarker data set obtained with the QUS in order to study the variation of these data in response to a rehabilitation intervention and to verify how these variations influence clinical data.

DETAILED DESCRIPTION:
A comprehensive clinical evaluation (questionnaires, clinical examination and ultrasound imaging) will be completed immediately before the intervention (pre), immediately after the intervention (post), and three months after the intervention (follow-up).

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with AT in the middle third of the Achilles tendon for at least six weeks
* AT signs objectified by the physical exam and the ultrasound imaging at the initial evaluation
* At least 18 years old
* Victorian Institute of Sport Assessment-Achilles Questionnaire (VISA-A) score below 90
* have pain of at least 3 out of 10 according to the analog visual scale during athletic activities

Exclusion Criteria:

* Pain at the Achilles tendon enthesis
* A complete rupture of the Achilles tendon History of Achilles tendon rupture Inflammatory arthropathy
* Sign of neurological lesion on physical examination of the lower limb
* Neurological disease (e.g. multiple sclerosis, stroke)
* History of intervention of the Achilles tendon or ankle (e.g. surgery, cortisone infiltration, extracorporeal shock waves therapy, platelet-rich plasma injection).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from patients with symptoms consistent with AT in the middle third of the Achilles tendon for at least six weeks. They will be recruited from physical therapy clinics, sports medicine clinic, sports teams and athletic clubs.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Responsiveness of a minimal data set of measures obtained with the QUS (quantitative ultrasonography) | 12 weeks
  The primary objective is to determine the responsiveness of a minimal data set of measures obtained with the QUS that characterize the biological integrity of the Achilles tendon (mean thickness, echogenicity, variance, homogeneity at 90 degrees, mean thickness, echogenicity and average homogeneity), after participants have completed the 12-week exercise program.

SECONDARY OUTCOMES:
Persistence of the QUS measures' modification at 3 months post-intervention | 12 weeks
  The second objective is to determine whether the immediate changes in the biological integrity of the tendon (pre vs post-intervention), characterized by the previous measures (mean thickness, echogenicity, variance, homogeneity at 90 degrees, mean thickness, echogenicity and average homogeneity), are maintained over time (three months post-intervention).

OTHER OUTCOMES:
Association between the QUS measures' modification and changes in the visual analog pain scale | 24 weeks
  The third objective is to verify whether the immediate and persistent changes are associated with changes in the visual analog pain scale, right after the 12-week exercise program and 12 weeks after the end of the exercise program. The visual analog pain scale is a pain scale that ranges from 0 to 10; 0 represents no pain and 10 represents an excruciating pain.
Association between the QUS measures' modification and changes in the Victorian Institute of Sports Assessment-Achilles questionnaire | 24 weeks
  The fourth objective is to verify whether the immediate and persistent changes are associated with changes in the Victorian Institute of Sports Assessment-Achilles questionnaire (VISA-A), right after the 12-week exercise program and 12 weeks after the end of the exercise program. The VISA-A score is a symptomatic scale that ranges from 0 and 100; 0 means that the participant is very symptomatic and 100 means the participant has no symptom.
Association between the QUS measures' modification and changes in the Lower Extremity Functional Scale | 24 weeks
  The fifth objective is to verify whether the immediate and persistent changes are associated with changes in the Lower Extremity Functional Scale (LEFS), right after the 12-week exercise program and 12 weeks after the end of the exercise program. The LEFS measures the functional impact of the pathology on the participant's daily life and it ranges from 0 to 80; 0 means that the Achilles tendinopathy has an extreme functional impact and 80 means it has no impact.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lamontagne, MD, Principal Investigator — Centre Hospitalier Universitaire de Montreal (CHUM)
Locations (1):
- Hôpital Hôtel-Dieu de Montreal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396
- [Result] Beyer R, Kongsgaard M, Hougs Kjaer B, Ohlenschlaeger T, Kjaer M, Magnusson SP. Heavy Slow Resistance Versus Eccentric Training as Treatment for Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1704-11. doi: 10.1177/0363546515584760. Epub 2015 May 27. PMID 26018970
- [Result] Binkley JM, Stratford PW, Lott SA, Riddle DL. The Lower Extremity Functional Scale (LEFS): scale development, measurement properties, and clinical application. North American Orthopaedic Rehabilitation Research Network. Phys Ther. 1999 Apr;79(4):371-83. PMID 10201543
- [Result] Cardoso TB, Pizzari T, Kinsella R, Hope D, Cook JL. Current trends in tendinopathy management. Best Pract Res Clin Rheumatol. 2019 Feb;33(1):122-140. doi: 10.1016/j.berh.2019.02.001. Epub 2019 Mar 8. PMID 31431267
- [Result] Collinger JL, Fullerton B, Impink BG, Koontz AM, Boninger ML. Validation of grayscale-based quantitative ultrasound in manual wheelchair users: relationship to established clinical measures of shoulder pathology. Am J Phys Med Rehabil. 2010 May;89(5):390-400. doi: 10.1097/PHM.0b013e3181d8a238. PMID 20407304
- [Result] de Jonge S, van den Berg C, de Vos RJ, van der Heide HJ, Weir A, Verhaar JA, Bierma-Zeinstra SM, Tol JL. Incidence of midportion Achilles tendinopathy in the general population. Br J Sports Med. 2011 Oct;45(13):1026-8. doi: 10.1136/bjsports-2011-090342. PMID 21926076
- [Result] Farnqvist K, Pearson S, Malliaras P. Adaptation of Tendon Structure and Function in Tendinopathy With Exercise and Its Relationship to Clinical Outcome. J Sport Rehabil. 2020 Jan 1;29(1):107-115. doi: 10.1123/jsr.2018-0353. PMID 30860421
- [Result] Kudron C, Carlson MJ, Meron A, Sridhar B, Brakke Holman R. Using Ultrasound Measurement of the Achilles Tendon in Asymptomatic Runners to Assist in Predicting Tendinopathy. J Ultrasound Med. 2020 Mar;39(3):491-496. doi: 10.1002/jum.15125. Epub 2019 Sep 6. PMID 31490583
- [Result] Lalumiere M, Lariviere C, Nadeau MJ, Paquette P, Lamontagne M, Desmeules F, Gagnon DH. Proposing a Minimal Data Set of Musculoskeletal Ultrasound Imaging Biomarkers to Inform Clinical Practice: An Analysis Founded on the Achilles Tendon. Ultrasound Med Biol. 2020 Sep;46(9):2222-2235. doi: 10.1016/j.ultrasmedbio.2020.04.024. Epub 2020 Jun 8. PMID 32527592
- [Result] McAuliffe S, Tabuena A, McCreesh K, O'Keeffe M, Hurley J, Comyns T, Purtill H, O'Neill S, O'Sullivan K. Altered Strength Profile in Achilles Tendinopathy: A Systematic Review and Meta-Analysis. J Athl Train. 2019 Aug;54(8):889-900. doi: 10.4085/1062-6050-43-18. Epub 2019 Aug 6. PMID 31386582
- [Result] Nadeau MJ, Desrochers A, Lamontagne M, Lariviere C, Gagnon DH. Quantitative ultrasound imaging of Achilles tendon integrity in symptomatic and asymptomatic individuals: reliability and minimal detectable change. J Foot Ankle Res. 2016 Aug 17;9:30. doi: 10.1186/s13047-016-0164-3. eCollection 2016. PMID 27540416
- [Result] Ortega-Avila AB, Reina-Martin I, Cervera-Garvi P, Lopezosa-Reca E, Cabello-Manrique D, Gijon-Nogueron G. Systematic review of the psychometric properties of the Victorian Institute of Sports Assessment - Achilles tendinopathy questionnaire. Disabil Rehabil. 2021 Apr;43(8):1056-1064. doi: 10.1080/09638288.2019.1652701. Epub 2019 Aug 20. PMID 31429326
- [Result] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Result] Wearing SC, Grigg NL, Hooper SL, Smeathers JE. Conditioning of the Achilles tendon via ankle exercise improves correlations between sonographic measures of tendon thickness and body anthropometry. J Appl Physiol (1985). 2011 May;110(5):1384-9. doi: 10.1152/japplphysiol.00075.2011. Epub 2011 Mar 10. PMID 21393469
- [Result] Rompe JD, Nafe B, Furia JP, Maffulli N. Eccentric loading, shock-wave treatment, or a wait-and-see policy for tendinopathy of the main body of tendo Achillis: a randomized controlled trial. Am J Sports Med. 2007 Mar;35(3):374-83. doi: 10.1177/0363546506295940. Epub 2007 Jan 23. PMID 17244902
- [Result] Sunding K, Fahlstrom M, Werner S, Forssblad M, Willberg L. Evaluation of Achilles and patellar tendinopathy with greyscale ultrasound and colour Doppler: using a four-grade scale. Knee Surg Sports Traumatol Arthrosc. 2016 Jun;24(6):1988-96. doi: 10.1007/s00167-014-3270-4. Epub 2014 Sep 6. PMID 25193569